CLINICAL TRIAL: NCT07007403
Title: The New Third Generation Video Laryngeal Mask Evaluation: a Pilot Study
Brief Title: The New Third Generation Video Laryngeal Mask Evaluation
Acronym: SACOVLM
Status: Completed | Type: Observational
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Principal Investigator, Michal Kalina, Deputy of medical director, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Other Study IDs: SACOVLM
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Supraglottic Airway
Keywords: supraglottic airway; laryngeal mask

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SaCo VLM laryngeal mask: In this group the video laryngeal mask is used for securing airway.

SUMMARY:
The goal of this study is to evaluate the performance of the new video laryngeal masks for securing airway in patients undergoing general anaesthesia. Main goal is to evaluate the first insertion attempt success rate, time to adequate ventilation, sealing pressures and adverse events.

DETAILED DESCRIPTION:
First, informed consent for study participation will be obtained from the patient. The consent will be collected during the preoperative evaluation by the anesthesiologist responsible for providing anesthesia care during the surgical procedure, in the preoperative holding area.

After obtaining informed consent, a routine preoperative assessment will be conducted by the anesthesiologist, including standard preparation procedures (e.g., establishing peripheral venous access, evaluation of airway management risk, etc.). Randomization will be performed using a computerized online tool (studyrandomizer.com).

The patient will then be transferred to the operating room, where standard monitoring will be initiated in accordance with the principles of safe anesthesia care.

Induction of anesthesia will follow, during which propofol and sufentanil will be administered in doses determined by the attending anesthesiologist. A muscle relaxant will not be used to facilitate insertion of the laryngeal mask airway (LMA). Once an adequate depth of anesthesia is achieved-defined by an entropy value of SE < 60-airway management will proceed according to the patient's assigned group (Group A - SaCoVLM; Group B - Supreme).

In both groups, the back of the LMA will be lubricated with a water-based gel. Group A will receive airway management using the SaCoVLM™ video laryngeal mask. Group B will receive airway management using the Supreme™ laryngeal mask.

The following data will be recorded: successful first attempt with adequate ventilation, time to initiation of ventilation, number of attempts required, SpO₂ at the time of ventilation onset, and EtCO₂ after initiation. Additionally, the fraction of oxygen in the exhaled gas mixture will be measured before the first insertion attempt and after achieving adequate ventilation. A gastric tube will be inserted via the drainage port in both groups.

Surgery will then proceed. During the procedure, oropharyngeal leak pressure will be measured at the 10th and 20th minute following LMA insertion. Ventilation will continue using the inserted LMA throughout the procedure. At the end of surgery, anesthesia will be discontinued, and the LMA will be removed. Upon removal, the presence of blood-tinged secretions on the LMA will be noted.

One hour after LMA removal, the patient will be assessed for oropharyngeal discomfort (e.g., sore throat, pain, cough irritation, or blood-streaked sputum). The need for oxygen therapy will also be recorded at 10 minutes and 1 hour following LMA removal. After this, the patient's participation in the study will conclude.

ELIGIBILITY:
Inclusion Criteria

* Patient without predicted difficult airway (MACOCHA score ≤ 2), undergoing a planned surgical procedure under general anesthesia with an indication for airway management using a laryngeal mask.
* Patient aged 18 years or older. Exclusion Criteria
* Patient younger than 18 years.
* Patient with predicted difficult airway (MACOCHA score > 2).
* Patient with a history of difficult airway.
* Patient requiring airway management with a method other than a laryngeal mask.
* Refusal or failure to sign the informed consent for study participation.
* Patient undergoing emergency surgery.
* Administration of muscle relaxants for LMA insertion.
* State Entropy value below 30 during LMA insertion.
* State Entropy value above 60 during LMA insertion.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing general anesthesia in the MNUL and Děčín Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-06-14 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
First insertion attempt success rate | From the start of the attempt to the end of the general anesthesia.
  First insertion attempt success rate. Successful attempt is considered if adequate ventilation is reached immediately after insertion without the need for realignment.

SECONDARY OUTCOMES:
Time to adequate ventilation | From the initiation of the first insertion attempt until the end of general anesthesia.
  Time from start of the insertion attempt until the adequate ventilation is reached. Adequate ventilation is considered if there are three or more plateau readings in EtCO2 curve.
Sealing pressure | From adequate ventilation until removing of the laryngeal mask.
  The maximum sealing pressure that can be reach after insertion and optimal alignment of the laryngeal mask. The APL ventilator will be set to 70 mbar and after there will be plateau on the pressure curve the sealing pressure will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Masarykova Nemocnice v Ústí nad Labem, Krajská Zdravotní a.s., Ústí nad Labem, Ústí Nad Labem Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided